CLINICAL TRIAL: NCT03444324
Title: A Randomized, Active-controlled, Multicenter, Phase III Study Investigating Efficacy and Safety of Intra-operative Use of BT524 (Human Fibrinogen Concentrate) in Subjects Undergoing Major Spinal or Abdominal Surgery (AdFIrst)
Brief Title: Adjusted Fibrinogen Replacement Strategy
Acronym: AdFIrst
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotest (Industry)
Collaborators: PRA Health Sciences (Industry); ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 995; 2017-001163-20 (EudraCT Number)
Record Dates: First submitted 2017-12-19; First posted 2018-02-23 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Bleeding Disorder; Hypofibrinogenemia; Acquired
Keywords: Fibrinogen
MeSH Terms: conditions — Hemostatic Disorders; Afibrinogenemia | interventions — cryoprecipitate coagulum

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to treatment with BT524 or FFP/Cryo.
Who Masked: Participant
Masking Description: Study 995 was partially blinded; surgeon, surgical staff and subjects were blinded to treatment allocation throughout the entire surgery. The subject was blinded throughout the study. The Investigational Medicinal Product (IMP), BT524 or FFP/Cryo, was administered by an unblinded anaesthesiologist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BT524 (Experimental): Investigational Human Fibrinogen Concentrate
  Interventions: Biological: BT524
- Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo) (Active Comparator): Standard of Care
  Interventions: Biological: FFP/Cryo

INTERVENTIONS:
Biological: BT524 — BT524 was administered intravenously at a patient specific dosage depending on the type of surgery, the extent of bleeding and the subject's clinical condition.
  Other Names: Human Fibrinogen concentrate
  Arms: BT524
Biological: FFP/Cryo — FFP/Cryo was administered intravenously; dosage according to local standards. FFP, 15 mL per kg body weight (BW); Cryoprecipitate, fixed dose of 10 units.
  Other Names: Fresh Frozen Plasma; Cryoprecipitate
  Arms: Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)

SUMMARY:
The main purpose of this study was to demonstrate the efficacy and safety of intraoperative use of fibrinogen concentrate BT524, as a complementary therapy for the management of uncontrolled severe hemorrhage in acquired hypofibrinogenemia. This non-inferiority study focused on the primary objective of demonstrating that BT524 is non-inferior that means not worse than the comparator fresh frozen plasma/cryoprecipitate in reducing intraoperative blood loss when administered intravenously in subjects with acquired hypofibrinogenemia undergoing elective major spinal or abdominal surgery.

DETAILED DESCRIPTION:
Fibrinogen is the first coagulation factor to become critically reduced during intraoperative bleeding. Therefore, rapid supplementation of fibrinogen to restore physiological plasma levels is an important component in achieving and maintaining hemostasis in bleeding patients. In this study, subjects with major blood loss during elective spinal surgery or abdominal surgery were randomized to receive either intravenous transfusion of the fibrinogen concentrate BT524, or fibrinogen-containing fresh frozen plasma/cryoprecipitate as first hemostatic intervention to rapidly replenish fibrinogen and control bleeding.

ELIGIBILITY:
Inclusion Criteria:

At screening:

1. Written informed consent
2. Subjects scheduled for elective major spinal surgery or cytoreductive pseudomyxoma peritonei (PMP) surgery with expected major blood loss
3. Male or female, aged ≥ 18 years
4. No increased bleeding risk as assessed by standard coagulation tests and medical history

Intra-operative:

5.

1. Subjects who underwent spinal surgery: Intra-operative clinically relevant bleeding of approximately 1 Liter, requiring hemostatic treatment during surgery.
2. Subjects who underwent cytoreductive PMP surgery: Intra-operative prediction of clinically relevant bleeding of more than 2 Liter, requiring hemostatic treatment during surgery

Exclusion Criteria:

1. Pregnancy or unreliable contraceptive measures or breast feeding (women only)
2. Hypersensitivity to proteins of human origin or known hypersensitivity reactions to components of the Investigational Medicinal Products (IMP)
3. Participation in another clinical study within 30 days before entering the study or during the study and/or previous participation in this study
4. Treatment with any fibrinogen concentrate and/or fibrinogen-containing product within 30 days prior to infusion of IMP
5. Employee or direct relative of an employee of the Contract Research Organization (CRO), the study site, or Biotest
6. Inability or lacking motivation to participate in the study
7. Medical condition, laboratory finding (e.g., clinically relevant biochemical or hematological findings outside the normal range), or physical exam finding that in the opinion of the investigator precludes participation
8. Presence or history of venous/arterial thrombosis or thromboembolic event (TEE) in the preceding 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niels Rahe-Meyer, Prof., Principal Investigator — Franziskus Hospital, Bielefeld
Locations (19):
- Belgium (2):
  - Site 02, Jette
  - Site 01, Leuven
- Czechia (4):
  - Site 54, Brno
  - Site 51, Prague
  - Site 53, Prague
  - Site 52, Ústí nad Labem
- Germany (5):
  - Site 15, Bielefeld
  - Site 11, Bonn
  - Site 12, Hanover
  - Site 14, München
  - Site 13, Münster
- Site 21, Warsaw, Poland
- Spain (4):
  - Site 31, Barcelona
  - Site 32, Barcelona
  - Site 33, Barcelona
  - Site34, Barcelona
- Switzerland (2):
  - Site 41, Liestal
  - Site 43, Zurich
- Site 71, Basingstoke, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahe-Meyer N, Roy A, Trouillier HH, Schimo S, Wessels-Kranz J, Abraha S, Staus A, Balaban U, Hader T, Schuttrumpf J, Aigner S, Bohm H. Efficacy and safety of human fibrinogen concentrate (BT524) in patients with major haemorrhage undergoing major orthopaedic or abdominal surgery (AdFIrst): a randomised, active-controlled, multicentre, partially blinded, phase 3 non-inferiority trial. EClinicalMedicine. 2025 Jun 7;85:103264. doi: 10.1016/j.eclinm.2025.103264. eCollection 2025 Jul. PMID 40741224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 339 subjects were screened, of these 222 subjects were eligible for the study and randomized. Baseline characteristics are available for the 222 randomized subjects.
Pre-assignment Details: There were 117 screen failures due to the following reasons: Eligibility criteria not met (before surgery), n=11; Intra-operative eligibility criterion not met, n=69; Physician decision, n=21; Adverse event, n=2; Withdrawal by subject, n=10; Technical reason, n=3; Other, n=1. Subjects eligible for randomization: n=222.
Groups:
- FFP/Cryo: Standard of Care
  Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo): FFP/Cryo was administered intravenously; dosage according to local standards. FFP, 15 mL per kg body weight (BW); Cryo, fixed dose of 10 units.
Period: Overall Study
Arm/Group | BT524 | FFP/Cryo
Started | 110 | 112
Completed | 105 | 106
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 4 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Trial Compliance | 1 | 1
Not completed — Physical disability to come to the site for the closing visit | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FFP/Cryo: Standard of Care
  Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo): FFP/Cryo was administered intravenously; dosage according to local standards. FFP, 15 mL per kg BW; Cryo, fixed dose of 10 units.
- Total: Total of all reporting groups
Arm/Group | BT524 | FFP/Cryo | Total
Number analyzed (Participants) | 110 | 112 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 58 | 120
  >=65 years | 48 | 54 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (12.52) | 60.8 (14.07) | 61.0 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 64 | 131
  Male | 43 | 48 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 103 | 106 | 209
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 109 | 107 | 216
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Czechia | 28 | 30 | 58
  Poland | 0 | 1 | 1
  United Kingdom | 48 | 50 | 98
  Switzerland | 9 | 9 | 18
  Germany | 14 | 9 | 23
  Spain | 11 | 13 | 24
Expected Blood Loss [Number; unit: participants]
  >1000 mL to <=2000 mL | 44 | 48 | 92
  >2000 mL | 66 | 64 | 130

OUTCOME MEASURES:

1. Primary Outcome: Intra-operative Blood Loss
Description: Intra-operative blood loss as measured by amount of blood from blood suction unit and amount of blood from surgical cloths and compresses.
Time Frame: From decision to treat the subject with IMP until end of surgery, an average of 5 hours
Population: Per-protocol set (PPS): All randomized subjects receiving IMP post randomization and with data collected post randomization. Subjects who were compliant with the trial protocol without any major protocol deviations thought to have the potential to impact the results of the efficacy analysis, e.g., no treatment or incomplete treatment with study intervention (BT524 or FFP/Cryo) during surgery, no postdose efficacy assessment for the primary endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Groups:
- Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo): Standard of Care
  Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo): FFP/Cryo was administered intravenously; dosage according to local standards.
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 103 | 98
mL | 1380.7 [1187.09 to 1574.31] | 1660.13 [1460.65 to 1859.61]
Statistical Analysis 1: Comparison: BT524 vs Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo); Test type: Non-Inferiority — The primary efficacy analysis of this endpoint was to test non-inferiority in the Per-protocol Set. The final analysis was performed using a two-way analysis of variance (ANOVA). Non-inferiority was to be demonstrated if the upper confidence limit of the two-sided 95 % confidence interval (CI) for the difference in the least squares mean (LSM) was less than the non-inferiority margin (150 mL); p < 0.001, Van Elteren test — p-value from Van Elteren test, stratified by predictive blood loss (> 1,000 mL to = 2,000 mL and >2,000 mL); Difference in LSM = -279.43, 95% CI 2-sided [-552.38 to -6.48]

2. Secondary Outcome: Proportion (%) of Subjects With Successful Correction of Fibrinogen Level (FIBTEM A10) 15 Minutes After Start of First IMP Administration
Description: Successful correction of the fibrinogen level is defined as restoring fibrinogen FIBTEM A10 baseline (prior surgery) levels measured by ROTEM (thromboelastometry) 15 minutes after start of first IMP administration
Time Frame: Prior first dose, 15 minutes after start of first IMP administration
Population: Modified Full Analysis Set (mFAS): All randomized subjects who received at least one dose of IMP prior to the 'end of surgery' and have at least one postdose efficacy assessment. This included all subjects whose IMP infusion started prior to the end of surgery, irrespective of the amount of IMP infused. Subjects were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo): Standard of Care
  FFP/Cryo: FFP/Cryo was administered intravenously; dosage according to local standards.
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 104 | 102
Participants | 59 | 19
Statistical Analysis 1: Comparison: BT524 vs Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; P-value is from a Cochran-Mantel-Haenszel model stratified by predictive blood loss (> 1,000 mL to ≤ 2,000 mL and > 2,000 mL); Difference in response rate = 38.1, 95% CI 2-sided [26 to 50.3]

3. Secondary Outcome: Time to First Successful Correction of Fibrinogen Level
Description: Correction of the fibrinogen level, measured via thromboelastometry (ROTEM/FIBTEM A10), within 15 minutes after IMP start, between 15 and 90 minutes after IMP start, after 90 minutes after IMP start, or unsuccessful correction. The 4 categories were compared between the two treatment arms using a Chi-square test.
Time Frame: prior 1st dose, pre-dose, 15 minutes and 90 minutes after start of first IMP administration, end of surgery
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 107 | 104
Participants
  <=15 minutes after IMP start | 59 | 19
  >15 and <= 90 minutes after IMP start | 17 | 11
  >90 minutes after IMP start | 11 | 16
  Unsuccessful correction | 20 | 58
Statistical Analysis 1: Comparison: BT524 vs Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo); Test type: Other; p < 0.001, Chi-squared

4. Secondary Outcome: Transfusion Requirements: Cell Salvage
Description: Total amount of transfusion products (allogeneic blood products) or autologous blood transfusion infused after start of first IMP administration until end of surgery. The end of surgery is defined as time of last suture.
Time Frame: After start of first IMP administration until end of surgery, an average of 5 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 107 | 104
mL | 95.6 (244.57) | 78.0 (234.77)

5. Secondary Outcome: Transfusion Requirements: Allogeneic Platelets
Description: as for outcome 4
Time Frame: After start of first IMP administration until end of surgery, an average of 5 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 107 | 104
mL | 3.0 (30.94) | 3.6 (36.38)

6. Secondary Outcome: Transfusion Requirements: Allogeneic Red Blood Cells
Description: as for outcome 4
Time Frame: After start of first IMP administration until end of surgery, an average of 5 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 107 | 104
mL | 455.5 (492.19) | 488.4 (547.72)

7. Secondary Outcome: Transfusion Requirements: Fresh Frozen Plasma
Description: as for outcome 4
Time Frame: After start of first IMP administration until end of surgery, an average of 5 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 107 | 104
mL | 60.5 (217.68) | 14.8 (110.94)

8. Secondary Outcome: Transfusion Requirements, Cryoprecipitate
Description: as for outcome 4
Time Frame: After start of first IMP administration until end of surgery, an average of 5 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 107 | 104
mL | 0 (0) | 0 (0)

9. Secondary Outcome: Amount of Red Blood Cells (RBCs)
Description: Amount (volume) of RBCs (allogenic and autologous RBCs) infused after start of first IMP administration until end of surgery. The end of surgery is defined as time of last suture.
Time Frame: After start of first IMP administration until end of surgery, an average of 5 hours
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 107 | 104
mL | 543.4 [441.99 to 644.77] | 558.9 [456.08 to 661.62]
Statistical Analysis 1: Comparison: BT524 vs Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo); Test type: Other; p < 0.831, ANOVA; Difference in LSM = -15.5, 95% CI 2-sided [-157.83 to 126.88]

10. Secondary Outcome: Post-operative Blood Loss
Description: Post-operative drainage volume in the first 24 hours after end of surgery
Time Frame: From end of surgery (time of last suture) up to 24 hours after the end of surgery
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 107 | 104
mL | 306.3 [234.15 to 378.38] | 293.9 [220.76 to 366.95]
Statistical Analysis 1: Comparison: BT524 vs Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo); Test type: Other; p = 0.809, ANOVA; Difference in LSM = 12.4, 95% CI 2-sided [-88.84 to 113.66]

11. Secondary Outcome: Subjects With Rebleeds
Description: Proportion (%) of subjects with rebleeds after the end of surgery until day 8
Time Frame: End of surgery up to 8 days after surgery
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 107 | 104
Participants | 0 | 5
Statistical Analysis 1: Comparison: BT524 vs Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo); Test type: Other; p = 0.022, Cochran-Mantel-Haenszel; Difference in proportion = -4.8, 95% CI 2-sided [-8.9 to -0.7]

12. Secondary Outcome: Hospital Length of Stay After Surgery
Description: Length of stay after surgery (days) = 'date of hospital discharge' minus 'date of surgery'. Where date of discharge is the date of discharge following the IMP treated surgery.
Time Frame: From day of surgery until day of hospital discharge, an average of 16 days (up to 56 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 107 | 104
Participants
  >36 days | 7 | 4
  29-36 days | 4 | 10
  22-28 days | 13 | 12
  15-21 days | 34 | 17
  8-14 days | 39 | 49
  1-7 days | 10 | 12

13. Secondary Outcome: In-hospital Mortality
Description: Number and percentages of subjects who died during hospital stay
Time Frame: From day of surgery until day of hospital discharge, an average of 16 days (up to 56 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 107 | 104
Participants | 0 | 0

14. Secondary Outcome: Number of Subjects With Thrombosis or Thromboembolic Events (TEEs)
Description: Total number of subjects with thrombosis or TEEs documented as treatment-emergent adverse events of special interest
Time Frame: From day of surgery until closing visit (up to 181 days)
Population: Safety Analysis Set (SAF): All subjects who have received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 110 | 112
Participants | 8 | 13

15. Secondary Outcome: Change in Viral Status
Description: Number of subjects with change in status of viral infections
Time Frame: Screening visit (up to 42 days prior to surgery) and closing visit (up to 181 days after surgery)
Population: Safety Analysis Set (SAF): All subjects who have received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
Number analyzed (Participants) | 110 | 112
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From day of surgery to closing visit (up to 181 days)
Description: Treatment emergent Adverse Events (TEAEs) defined as any Adverse Events (AEs) with start during or after administration of Investigational Medicinal Product (IMP) until the subject's last trial visit. Non-TEAEs defined as any AEs after signing the Informed Consent Form (ICF) and prior administration of IMP. Analyses were focused on TEAEs.
Arm/Group | BT524 | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo)
All-Cause Mortality (participants affected / at risk) | 0/110 | 1/112
Serious Adverse Events (participants affected / at risk) | 28/110 | 41/112
Other Adverse Events (participants affected / at risk) | 92/110 | 93/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT524 (N=110) | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo) (N=112)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (3)
Neurogenic shock (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 2 (2) | 1 (1) — General disorders and administration site conditions
Chest pain (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Pain (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Surgical failure (General disorders) | 0 (0) | 1 (1) — General disorders and administration site conditions
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Dural tear (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Bladder injuryI (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 2 (2) | 0 (0)
Paraparesis (Nervous system disorders) | 2 (2) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 3 (3)
Wound infection (Infections and infestations) | 1 (1) | 2 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT524 (N=110) | Fresh Frozen Plasma (FFP)/Cryoprecipitate (Cryo) (N=112)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 8 (8)
Oxygen saturation decreased (Investigations) | 2 (2) | 7 (8)
Anaemia postoperative (Injury, poisoning and procedural complications) | 15 (15) | 6 (6)
Hypotension (Vascular disorders) | 23 (29) | 10 (14)
Tachycardia (Cardiac disorders) | 19 (22) | 14 (14)
Constipation (Gastrointestinal disorders) | 6 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (11) | 4 (4)
Hypertransaminasaemia (Hepatobiliary disorders) | 13 (13) | 11 (11)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6)
Hallucination (Psychiatric disorders) | 29 (30) | 26 (26)
Pneumonia (Infections and infestations) | 10 (10) | 10 (10)
Urinary tract infection (Infections and infestations) | 10 (10) | 10 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol: 995_Protocol_V4.0 (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT03444324/Prot_000.pdf
  • Study Protocol: 995_Protocol_V4.3_UK (2021-09-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT03444324/Prot_001.pdf
  • Statistical Analysis Plan (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT03444324/SAP_002.pdf
  • Informed Consent Form (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03444324/ICF_003.pdf